CLINICAL TRIAL: NCT01813916
Title: Identification and Characterization of the Biomarker in Synovial Fluid for Hyaluronic Acid Therapy in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 200804039R
Record Dates: First submitted 2013-01-30; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; synovial fluid; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- proteomic analysis (No Intervention)
  Interventions: Other: proteomic analysis

INTERVENTIONS:
Other: proteomic analysis

SUMMARY:
The purpose of this study is to use the proteomic analysis of synovial fluid to perform the comprehensive investigation of the biomarker that will be useful to assign the tratment effectiveness of five weekly intra-articular HA injection.

DETAILED DESCRIPTION:
The intra-articular injection with HA is an accepted therapy for OA. However, the exact regulation of HA treatment is unclear. Compared the expression SF proteome from OA patients who received HA/800 treatment or not (post and pre-HA treatment) may be possible to identify the protein that response to the HA treatment and apply this to prognosis of OA. We used two-dimensional difference gel electrophoresis (2D-DIGE) combined with matrix-assisted laser desorption ionization time of light mass spectrometry (MALDI-TOF) to determine the differentially displayed proteins in human SF. Finally, we used Western blotting and ELISA analysis to validate the potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis
* Accept the intra-articular HA injection therapy

Exclusion Criteria:

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To study the protein expression of synovial fluid for hyaluronic acid therapy in osteoarthritis | up to 12 months
  We used two-dimensional difference gel electrophoresis (2D-DIGE) combined with matrix-assisted laser desorption ionization time of light mass spectrometry (MALDI-TOF) to determine the differentially displayed proteins in human synovial fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chuan Jiang, M.D.;Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Ccj@Ntu.Edu.Tw, Taipei, Taiwan